CLINICAL TRIAL: NCT06028126
Title: Efficacy of Intermittent Superficial Parasternal Intercostal Plane Block on Postoperative Pain Control in Patients Undergoing Cardiac Surgery With Median Sternotomy - EPOCH Randomized Clinical Trial
Brief Title: Superficial Parasternal Intercostal Plane Block in Cardiac Surgery Trial
Acronym: EPOCH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Queen Elizabeth II Health Sciences Centre (Other); Foothills Medical Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23-038
Record Dates: First submitted 2023-08-08; First posted 2023-09-08 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-10

CONDITIONS: Post-operative Pain; Post-operative Delirium; Post-cardiac Surgery; Chronic Pain; Opioid Use Disorder; Anesthesia, Local
MeSH Terms: conditions — Pain, Postoperative; Emergence Delirium; Chronic Pain; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The patient, intervention appliers (i.e. the operating room staff), medical practitioners, and outcome assessors will all be blinded to the randomized treatment arm until the database is locked. Unblinding procedures will be made available for breaking codes if necessary for clinical treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.2% ropivacaine (Experimental): Intermittent superficial parasternal intercostal plane block via ultrasound-guided catheter placement. Initial bolus dosing of 20 milliliter (mL) of 0.2% ropivacaine per side at the time of catheter placement, followed by intermittent boluses of 10 mL 0.2% ropivacaine per side.
  Interventions: Procedure: Intermittent Superficial Parasternal Intercostal Plane Block - Experimental
- 0.9% saline (Sham Comparator): Intermitted superficial parasternal intercostal plane block via ultrasound-guided catheter placement. Initial bolus of 20 mL of 0.9% saline per side at the time of catheter placement, followed by intermitted boluses of 10 ml of 0.9% saline per side.
  Interventions: Procedure: Intermittent Superficial Parasternal Intercostal Plane Block - Sham

INTERVENTIONS:
Procedure: Intermittent Superficial Parasternal Intercostal Plane Block - Experimental — Catheter insertion will be performed by an anesthesiologist with regional block training immediately following skin closure in the operating room. Catheters will be inserted under ultrasound guidance, in a sterile fashion, with a high-frequency linear transducer which will be placed 1 cm lateral to the sternal border in the longitudinal plane in order to view the T4-T5 intercostal space. A Tuohy needle will be used to enter the superficial parasternal intercostal plane, with saline being injected to help visualize the plane between the pectoralis major and intercostal muscles. Subsequently, the catheters will be advanced into the plane, and secured on the skin.
  Following initial bolus dosing at the time of catheter placement (20 mL 0.2% ropivacaine), intermittent boluses of 10 mL 0.2% ropivacaine per side will be delivered via catheters q6-8 hours for 48 hours post-catheter insertion.
  Arms: 0.2% ropivacaine
Procedure: Intermittent Superficial Parasternal Intercostal Plane Block - Sham — Catheter insertion will be performed by an anesthesiologist with regional block training immediately following skin closure in the operating room. Catheters will be inserted under ultrasound guidance, in a sterile fashion, with a high-frequency linear transducer which will be placed 1 cm lateral to the sternal border in the longitudinal plane in order to view the T4-T5 intercostal space. A Tuohy needle will be used to enter the superficial parasternal intercostal plane, with saline being injected to help visualize the plane between the pectoralis major and intercostal muscles. Subsequently, the catheters will be advanced into the plane, and secured on the skin.
  Following initial bolus dosing at the time of catheter placement (20 mL 0.9% Saline), intermittent boluses of 10 mL 0.9% Saline per side will be delivered via catheters q6-8 hours for 48 hours post-catheter insertion.
  Arms: 0.9% saline

SUMMARY:
The goal of this clinical trial is to assess whether the use of intermittent superficial parasternal intercostal plane blocks reduces opioid usage in patients undergoing cardiac surgery with median sternotomy.

Participants randomized to the intervention group will receive the blocks with 0.2% ropivacaine administered via catheters placed in the superficial parasternal intercostal plane bilaterally under ultrasound guidance. Researchers will compare this group with a control group given 0.9% saline through similarly placed catheters. The primary outcome will be cumulative postoperative opioid use (measured as Milligram Morphine Equivalent (MME)) up to 72 hours following catheter insertion.

DETAILED DESCRIPTION:
This trial is comparing the use of 0.2% ropivacaine and 0.9% saline through a parasternal intercostal plane block and to measure whether there are any tangible changes in:

1. The primary outcome will be cumulative postoperative opioid use (measured as Milligram Morphine Equivalent (MME)) up to 72 hours following catheter insertion.

   Secondary outcomes will be:
2. cumulative postoperative opioid use from catheter insertion up to hospital discharge - measured as MME
3. median pain score - measured at rest and with coughing using a standardized numerical rating scale - for 72 hours post catheter insertion
4. delirium - assessed twice daily using institutional scores up to 72 hours following catheter insertion.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgery via median sternotomy

Exclusion Criteria:

* Redo sternotomy, or cardiac surgery performed through non-sternotomy approaches (minimally invasive procedures, thoracotomies, mini-sternotomy, hemi-sternotomy, etc.)
* Emergency procedures (surgery within 2 hours)
* Clinical instability which in the judgement of the investigator precludes enrollment or participation in the study
* Weight < 50kg
* Active systemic bacterial infection including infective endocarditis or pre-existing sternal infections
* Surgery for infective endocarditis
* Pregnancy or nursing
* Chronic opioid/narcotic use > 6 weeks, active use of illicit drugs, long-term opioid exposure or chronic pain disorder/syndromes
* Allergies to amide anesthetic agents or any components of study interventions
* Inability to comply with, or participate in, protocol (i.e. cognitive impairment/altered mental status/neurological deficit or disorder, inability to provide informed consent, inability to complete pain rating scales, etc.)
* Receipt of an investigational drug or device within past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative postoperative opioid use up to 72 hours | 72 hours after catheter insertion.
  Postoperative opioid use measured using Milligram Morphine Equivalent(MME) from catheter insertion up to 72 hours.

SECONDARY OUTCOMES:
Median pain score | over 72 hours post-extubation
  Measured using visual analog pain scale (minimum 0, maximum 10; higher is worse)
Cumulative post-operative opioid use | from time of catheter insertion until discharge from hospital
  Opioid use measured using MME
Delirium | for 72 hours following catheter insertion
  assessed using Confusion Assessment Method (positive or negative; positive indicates delirium present) or Intensive Care Unit Delirium Screen Checklist Score (minimum 0, maximum 8; higher scores is worse; score greater than 3 is positive for delirium) or more than one dose antipsychotic drug or clinical diagnosis by psychiatrist.
Quality of Recovery-15 Scale | 24-96 hours post surgery
  Assessed using Quality of Recovery-15 Scale (minimum 0, maximum 150; higher scores mean a better outcome)

OTHER OUTCOMES:
Time from catheter insertion to extubation | from time of catheter insertion until extubation
  Measured time from catheter insertion to extubation
Time from catheter insertion to first analgesic request | immediately after the intervention
  Measured time from catheter insertion to first analgesic request
Time from catheter insertion to mobilization | From the time of catheter insertion to mobilization
  Measured time from catheter insertion to mobilization
ICU and hospital length of stay | From date of surgery until date of ICU and Hospital discharge
  Measured time of ICU and hospital length of stay
Postoperative nausea and vomiting | Up to 72 hours following catheter insertion
  Measured via a 10-point visual analogue scale (minimum 0, maximum 10; higher scores are worse)
Quality of Recovery-15 Scale | Post-operative day 4-7
  Assessed using Quality of Recovery-15 Scale (minimum: 0, maximum: 150; higher scores mean a better outcome)
Post thoracotomy Pain | Assessed at 3 months +/- 4 weeks
  Assessed using McGill Pain Questionnaire (minimum 0, maximum 78; higher scores mean a worse outcome) and Patient-Reported Outcomes Measurement Information System 29-Item Profile (PROMIS 29) Subsections:
  Physical Function: 4-20, higher scores is better outcome. Anxiety: 4-20, higher scores is worse outcome. Depression: 4-20, higher scores is worse outcome. Fatigue: 4-20, higher scores is worse outcome. Sleep Disturbance: 4-20, higher scores is worse outcome. Ability to Participate in Social Roles and Activities: 4-20, higher scores is better outcome.
  Pain Interference: 4-20, higher scores is worse outcome. Pain Intensity: 0-10 higher scores is worse outcome.)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Alli, MD, Principal Investigator — Unity Health Toronto
Locations (4):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Royal Columbian Hospital, Vancouver, British Columbia
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mueller XM, Tinguely F, Tevaearai HT, Revelly JP, Chiolero R, von Segesser LK. Pain location, distribution, and intensity after cardiac surgery. Chest. 2000 Aug;118(2):391-6. doi: 10.1378/chest.118.2.391. PMID 10936130
- [Background] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Background] Zhang Y, Min J, Chen S. Continuous Pecto-Intercostal Fascial Block Provides Effective Analgesia in Patients Undergoing Open Cardiac Surgery: A Randomized Controlled Trial. Pain Med. 2022 Mar 2;23(3):440-447. doi: 10.1093/pm/pnab291. PMID 34601602
- [Background] Dost B, De Cassai A, Balzani E, Tulgar S, Ahiskalioglu A. Effects of ultrasound-guided regional anesthesia in cardiac surgery: a systematic review and network meta-analysis. BMC Anesthesiol. 2022 Dec 29;22(1):409. doi: 10.1186/s12871-022-01952-7. PMID 36581838
- [Background] Kumar AK, Chauhan S, Bhoi D, Kaushal B. Pectointercostal Fascial Block (PIFB) as a Novel Technique for Postoperative Pain Management in Patients Undergoing Cardiac Surgery. J Cardiothorac Vasc Anesth. 2021 Jan;35(1):116-122. doi: 10.1053/j.jvca.2020.07.074. Epub 2020 Jul 30. PMID 32859487
- [Background] Brown CR, Chen Z, Khurshan F, Groeneveld PW, Desai ND. Development of Persistent Opioid Use After Cardiac Surgery. JAMA Cardiol. 2020 Aug 1;5(8):889-896. doi: 10.1001/jamacardio.2020.1445. PMID 32584934
- [Background] Barletta JF. Clinical and economic burden of opioid use for postsurgical pain: focus on ventilatory impairment and ileus. Pharmacotherapy. 2012 Sep;32(9 Suppl):12S-8S. doi: 10.1002/j.1875-9114.2012.01178.x. PMID 22956490
- [Background] Bovill JG, Sebel PS, Stanley TH. Opioid analgesics in anesthesia: with special reference to their use in cardiovascular anesthesia. Anesthesiology. 1984 Dec;61(6):731-55. PMID 6150663
- [Background] Gan TJ. Poorly controlled postoperative pain: prevalence, consequences, and prevention. J Pain Res. 2017 Sep 25;10:2287-2298. doi: 10.2147/JPR.S144066. eCollection 2017. PMID 29026331